CLINICAL TRIAL: NCT01764815
Title: Evaluation of Directional Stimulation During the Implantation of Deep Brain Stimulation Leads for the Treatment of Movement Disorders
Brief Title: Evaluation of Directional Stimulation During the Implantation of Deep Brain Stimulation (DBS) Leads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aleva Neurotherapeutics SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KEK 072-12; CIV-12-08-008482 (Other: EUDAMED)
Record Dates: First submitted 2012-12-26; First posted 2013-01-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Parkinson's Disease; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Directional lead (Experimental)
  Interventions: Device: directSTN Acute lead connected to external neurostimulator

INTERVENTIONS:
Device: directSTN Acute lead connected to external neurostimulator — Test phase will be performed intra-operatively, prior to chronic lead implant

SUMMARY:
The purpose of this study is to provide proof-of-concept that directional stimulation, in an intraoperative setting, is perceivable in a subject and is different from omnidirectional stimulation. The tests will be performed using a dedicated DBS lead connected to external neurostimulator.

ELIGIBILITY:
Inclusion Criteria:

* Subject is indicated to undergo DBS for Parkinson's disease or Essential Tremor according to criteria of the Study site
* For Parkinson Disease:

  * Person is between 18 and 75 years of age
  * Established diagnosis of idiopathic Parkinson's disease with progression of symptoms for a minimum of 2 years.
  * Person has a history of at least 30% improvement on the Unified Parkinson's Disease Rating Scale with therapy in L-dopa (levodopa)
  * Weak control of symptoms by dopaminergic therapy (off phenomenon, fluctuations on / off, dyskinesia on)
* For Essential Tremor:

  * Person is between 18 and 80 years of age
  * Established diagnosis of Essential Tremor for a minimum of 2 years
  * Functional disability due to tremor was not adequately controlled by medication for at least 3 months prior to implant.
* Person has given his/her written consent

Exclusion Criteria:

* Person suffering from an active major psychiatric disorder
* Mattis Dementia Rating Scale score <130 or otherwise not capable of discernment
* Presence of major co-morbidity or medical condition that may affect participation to the study
* Presence of an electrical or electromagnetic implant (e.g., cochlear implant, pacemaker)
* Person with a previous surgery for the treatment of Parkinson's disease or Essential Tremor
* Person with a previous brain ablation procedure
* Person who suffers from epilepsy
* Person who is pregnant: a pregnancy test will be performed in women of childbearing age
* Person with coagulopathies
* Abuse of drugs or alcohol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Measurement of the therapeutic window's boundaries when stimulating in specific angular directions, and comparison to those obtained when stimulating in all directions. | up to one hour during surgery
  A therapeutic window is defined as the difference between the electrical current threshold at which a desired therapeutic effect is obtained and the current threshold at which side effects appear.

SECONDARY OUTCOMES:
Electrical functionality of the study device during the test phase | 1 day
  The electrical integrity of the device will be measured before and after its use, to confirm that it was functional throughout the test phase.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Pollo, PD, Dr. med, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Inselspital University Hospital, Bern, Switzerland